CLINICAL TRIAL: NCT00330213
Title: Effects of Red Wine and Cognac on Coronary Circulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Tampere University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KLF-RW-06
Record Dates: First submitted 2006-05-24; First posted 2006-05-26 (Estimated); Last update posted 2006-05-26 (Estimated); Status verified 2004-09

CONDITIONS: Healthy
Keywords: transthoracic; echocardiography; red wine; cognac; coronary reactivity

INTERVENTIONS:
Behavioral: red wine and cognac consumption

SUMMARY:
Red wine consumption is associated with reduced cardiovascular disease mortality, and the cardioprotective properties may be partly related to its ability to improve endothelial function. The purpose of this study was to determine whether moderate doses of red wine, de-alcoholized red wine and cognac improve coronary flow reserve.

DETAILED DESCRIPTION:
Moderate consumption of red wine is associated with reduced coronary artery disease mortality. Cardioprotective effects of red wine may be partly related to its ability to improve endothelial function. Red wine increases endothelium-dependent flow-mediated dilatation of the brachial artery acutely after ingestion. Moreover, a heavy dose of red wine (ethanol 1.0 g/kg) has been shown to increase coronary flow reserve (CFR) as measured with transthoracic Doppler echocardiography. CFR depicts the relative increase of coronary blood flow in response to maximal myocardial hyperemia induced by adenosine. It is reduced in atherosclerosis and various conditions associated with the dysfunction of coronary microcirculation, such as diabetes and hypercholesterolemia.

Both ethanol and antioxidative polyphenols have been implicated in beneficial endothelial effects of red wine. However, their relative contributions remain uncertain in vivo. It has been suggested that red wine has stronger vasoactive properties than other alcohol beverages, and even de-alcoholized red wine may be sufficient to improve flow-mediated dilatation of the brachial artery. Cognac is also known to contain polyphenols, but its effects on coronary circulation have not been evaluated.

The purpose of this randomized controlled cross-over study was to determine with transthoracic echocardiography whether moderate doses of red wine improve CFR in response to adenosine in healthy humans. We also studied contributions of ethanol and antioxidants by comparing the effects of equal doses of alcoholic and de-alcoholized red wine, and cognac on the plasma antioxidant capacity and CFR.

ELIGIBILITY:
Inclusion Criteria:

* healthy males

Exclusion Criteria:

* smoking, medication of any kind

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2004-10; Study Completion 2005-04

PRIMARY OUTCOMES:
coronary flow reserve
plasma antioxidant capacity

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas O Kiviniemi, MD, Principal Investigator — Dept. Clinical Physiology and Nuclear Medicine, Turku University Hospital
Locations (1):
- Dept. Clinical Physiology and Nuclear Medicine, Turku University Hospital, Turku, Finland

REFERENCES:
- [Background] Kiviniemi TO, Saraste M, Koskenvuo JW, Airaksinen KE, Toikka JO, Saraste A, Parkka JP, Hartiala JJ. Coronary artery diameter can be assessed reliably with transthoracic echocardiography. Am J Physiol Heart Circ Physiol. 2004 Apr;286(4):H1515-20. doi: 10.1152/ajpheart.00819.2003. Epub 2003 Dec 4. PMID 14656707
- [Derived] Kiviniemi TO, Saraste A, Toikka JO, Saraste M, Raitakari OT, Parkka JP, Lehtimaki T, Hartiala JJ, Viikari J, Koskenvuo JW. Effects of cognac on coronary flow reserve and plasma antioxidant status in healthy young men. Cardiovasc Ultrasound. 2008 Jun 3;6:25. doi: 10.1186/1476-7120-6-25. PMID 18522727